CLINICAL TRIAL: NCT03676010
Title: Definition for the Assessment of Time-to-event Endpoints in CANcer Trials (DATECAN-1) : Formal Consensus Method for the Development of Guidelines for Standardized Time-to-event Endpoints' Definitions in Cancer Clinical Trials
Brief Title: Definition for the Assessment of Time-to-event Endpoints in CANcer Trials (DATECAN-1)
Acronym: DATECAN-1
Status: Active, not recruiting | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government); Institut du Cancer de Montpellier - Val d'Aurelle (Other); Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: IB2009-DATECAN-1
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Cancer; Randomized controlled trial; Endpoint; Consensus
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Sarcoma and GIST: Experts involved in the consensus process for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for patients with Sarcoma and GIST
  Interventions: Other: Sarcoma and GIST
- Breast cancer: Experts involved in the consensus process for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for patients with Breast cancer
  Interventions: Other: Breast cancer
- Pancreatic cancer: Experts involved in the consensus process for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for patients with Pancreatic cancer
  Interventions: Other: Pancreatic cancer
- Renal cell carcinoma: Experts involved in the consensus process for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for patients with Renal cell carcinoma
  Interventions: Other: Renal cell carcinoma
- Colon Cancer (adjuvant setting): Experts involved in the consensus process for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for patients with Colon Cancer (adjuvant setting)
  Interventions: Other: Colon cancer
- Solid tumours undergoing image-guided tumor ablation: Experts involved in the consensus process for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for patients with Solid tumours undergoing image-guided tumor ablation
  Interventions: Other: Solid tumours undergoing image-guided tumor ablation
- (early) Non Small Cell Lung Cancer: Experts involved in the consensus process for providing recommandations for the definitions of time to event outcomes to be used in randomized trials for patients with (early) Non Small Cell Lung Cancer
  Interventions: Other: (early) Non Small Cell Lung Cancer

INTERVENTIONS:
Other: Sarcoma and GIST — No Intervention : Consensus of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.
  Groups: Sarcoma and GIST
Other: Breast cancer — No intervention : Consensus of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.
  Groups: Breast cancer
Other: Pancreatic cancer — No intervention : Consensus of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.
  Groups: Pancreatic cancer
Other: Renal cell carcinoma — No intervention : Consensus of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.
  Groups: Renal cell carcinoma
Other: Colon cancer — No intervention : Consensus of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy (adjuvant setting).
  Groups: Colon Cancer (adjuvant setting)
Other: Solid tumours undergoing image-guided tumor ablation — No intervention : Consensus of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.
  Groups: Solid tumours undergoing image-guided tumor ablation
Other: (early) Non Small Cell Lung Cancer — No intervention : Consensus of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.
  Groups: (early) Non Small Cell Lung Cancer

SUMMARY:
In randomised phase III cancer clinical trials, the most objectively defined and only validated time-to-event endpoint is overall survival (OS). The appearance of new types of treatments and the multiplication of lines of treatment have resulted in the use of surrogate endpoints for overall survival such as progression-free survival (PFS), or time-to-treatment failure. Their development is strongly influenced by the necessity of reducing clinical trial duration, cost and number of patients. However, while these endpoints are frequently used, they are often poorly defined and definitions can differ between trials which may limit their use as primary endpoints. Moreover, this variability of definitions can impact on the trial's results by affecting estimation of treatments' effects. The aim of the Definition for the Assessment of Time-to-event Endpoints in CANcer trials (DATECAN) project is to provide recommendations for standardised definitions of time-to-event endpoints in randomised cancer clinical trials.

We will use a formal consensus methodology based on experts' opinions which will be obtained in a systematic manner.

Definitions will be independently developed for several cancer sites, including pancreatic, breast, head and neck and colon cancer, as well as sarcomas and gastrointestinal stromal tumours (GISTs).

The DATECAN project should lead to the elaboration of recommendations that can then be used as guidelines by researchers participating in clinical trials. This process should lead to a standardisation of the definitions of commonly used time-to-event endpoints, enabling appropriate comparisons of future trials' results.

DETAILED DESCRIPTION:
There is no methodology to provide appropriate definitions for survival endpoints. As such, including or excluding an event in a survival endpoint definition is only based on opinion from experts. For this reason, we launched the DATECAN-1 project in 2009. Its objective is to elaborate standardized definitions for survival endpoints in randomized clinical trials, based on a rigorous and validated consensus methodology. Once this project will be finalized (2012), guidelines for the definitions of survival endpoints to be used in clinical trials will be available.

This collaborative work involves the network of the statisticians from Regional Comprehensive Cancer Centers (Bordeaux, Lille, Montpellier, Dijon, Paris, Toulouse), the network of the Cancer Data Centers (CTD) of the French National Cancer Institute (INCA; Montpellier, Bordeaux, Curie, Dijon-GERCOR) as well as the Headquarters from the European Organization for Research and Treatment of Cancer (EORTC). This project is supported by a 2009 grant from the French League Against Cancer .

The DATECAN-1 project relies on a validated formal consensus method (Fitch K. The Rand/UCLA appropriateness method user's manual. 2001). This consensus approach formalizes the degree of agreement among experts by identifying and selecting the points on which experts agree, disagree or are undecided. The guidelines are subsequently based on agreement points. It is a rigorous and explicit method since it involves international experts in clinical trials in the field of the targeted cancer localizations. This method involves two rounds of rating (questionnaires) and an in-person meeting to address points for which consensus has not been reached yet.

We published the methodology of the consensus process (Bellera et al. Eur J Cancer 2013).

Guidelines have now been published following the international consensus process, for pancreatic cancer, sarcoma and GIST, beast cancer and renal cell carcinoma (See "Citations filed" below). For other localization (head and neck, stomach, colon): guidelines are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Sarcoma / GIST
* Breast cancer
* Pancreatic cancer
* Renal cell carcinoma
* adjuvant colon cancer
* early non small cell lung cancer

Exclusion Criteria :

- Individual patient data unavailable

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No patient will be included.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Institut du Cancer de Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puijk RS, Ahmed M, Adam A, Arai Y, Arellano R, de Baere T, Bale R, Bellera C, Binkert CA, Brace CL, Breen DJ, Brountzos E, Callstrom MR, Carrafiello G, Chapiro J, de Cobelli F, Coupe VMH, Crocetti L, Denys A, Dupuy DE, Erinjeri JP, Filippiadis D, Gangi A, Gervais DA, Gillams AR, Greene T, Guiu B, Helmberger T, Iezzi R, Kang TW, Kelekis A, Kim HS, Kroncke T, Kwan S, Lee MW, Lee FT, Lee EW Jr, Liang P, Lissenberg-Witte BI, Lu DS, Madoff DC, Mauri G, Meloni MF, Morgan R, Nadolski G, Narayanan G, Newton I, Nikolic B, Orsi F, Pereira PL, Pua U, Rhim H, Ricke J, Rilling W, Salem R, Scheffer HJ, Sofocleous CT, Solbiati LA, Solomon SB, Soulen MC, Sze D, Uberoi R, Vogl TJ, Wang DS, Wood BJ, Goldberg SN, Meijerink MR. Consensus Guidelines for the Definition of Time-to-Event End Points in Image-guided Tumor Ablation: Results of the SIO and DATECAN Initiative. Radiology. 2021 Dec;301(3):533-540. doi: 10.1148/radiol.2021203715. Epub 2021 Sep 28. PMID 34581627
- [Result] Bellera CA, Penel N, Ouali M, Bonvalot S, Casali PG, Nielsen OS, Delannes M, Litiere S, Bonnetain F, Dabakuyo TS, Benjamin RS, Blay JY, Bui BN, Collin F, Delaney TF, Duffaud F, Filleron T, Fiore M, Gelderblom H, George S, Grimer R, Grosclaude P, Gronchi A, Haas R, Hohenberger P, Issels R, Italiano A, Jooste V, Krarup-Hansen A, Le Pechoux C, Mussi C, Oberlin O, Patel S, Piperno-Neumann S, Raut C, Ray-Coquard I, Rutkowski P, Schuetze S, Sleijfer S, Stoeckle E, Van Glabbeke M, Woll P, Gourgou-Bourgade S, Mathoulin-Pelissier S. Guidelines for time-to-event end point definitions in sarcomas and gastrointestinal stromal tumors (GIST) trials: results of the DATECAN initiative (Definition for the Assessment of Time-to-event Endpoints in CANcer trials)dagger. Ann Oncol. 2015 May;26(5):865-872. doi: 10.1093/annonc/mdu360. Epub 2014 Jul 28. PMID 25070543
- [Result] Bonnetain F, Bonsing B, Conroy T, Dousseau A, Glimelius B, Haustermans K, Lacaine F, Van Laethem JL, Aparicio T, Aust D, Bassi C, Berger V, Chamorey E, Chibaudel B, Dahan L, De Gramont A, Delpero JR, Dervenis C, Ducreux M, Gal J, Gerber E, Ghaneh P, Hammel P, Hendlisz A, Jooste V, Labianca R, Latouche A, Lutz M, Macarulla T, Malka D, Mauer M, Mitry E, Neoptolemos J, Pessaux P, Sauvanet A, Tabernero J, Taieb J, van Tienhoven G, Gourgou-Bourgade S, Bellera C, Mathoulin-Pelissier S, Collette L. Guidelines for time-to-event end-point definitions in trials for pancreatic cancer. Results of the DATECAN initiative (Definition for the Assessment of Time-to-event End-points in CANcer trials). Eur J Cancer. 2014 Nov;50(17):2983-93. doi: 10.1016/j.ejca.2014.07.011. Epub 2014 Sep 22. PMID 25256896
- [Result] Bellera CA, Pulido M, Gourgou S, Collette L, Doussau A, Kramar A, Dabakuyo TS, Ouali M, Auperin A, Filleron T, Fortpied C, Le Tourneau C, Paoletti X, Mauer M, Mathoulin-Pelissier S, Bonnetain F. Protocol of the Definition for the Assessment of Time-to-event Endpoints in CANcer trials (DATECAN) project: formal consensus method for the development of guidelines for standardised time-to-event endpoints' definitions in cancer clinical trials. Eur J Cancer. 2013 Mar;49(4):769-81. doi: 10.1016/j.ejca.2012.09.035. Epub 2012 Nov 2. PMID 23122780
- [Result] Gourgou-Bourgade S, Cameron D, Poortmans P, Asselain B, Azria D, Cardoso F, A'Hern R, Bliss J, Bogaerts J, Bonnefoi H, Brain E, Cardoso MJ, Chibaudel B, Coleman R, Cufer T, Dal Lago L, Dalenc F, De Azambuja E, Debled M, Delaloge S, Filleron T, Gligorov J, Gutowski M, Jacot W, Kirkove C, MacGrogan G, Michiels S, Negreiros I, Offersen BV, Penault Llorca F, Pruneri G, Roche H, Russell NS, Schmitt F, Servent V, Thurlimann B, Untch M, van der Hage JA, van Tienhoven G, Wildiers H, Yarnold J, Bonnetain F, Mathoulin-Pelissier S, Bellera C, Dabakuyo-Yonli TS. Guidelines for time-to-event end point definitions in breast cancer trials: results of the DATECAN initiative (Definition for the Assessment of Time-to-event Endpoints in CANcer trials). Ann Oncol. 2015 Dec;26(12):2505-6. doi: 10.1093/annonc/mdv478. Epub 2015 Oct 13. No abstract available. PMID 26467471
- [Result] Kramar A, Negrier S, Sylvester R, Joniau S, Mulders P, Powles T, Bex A, Bonnetain F, Bossi A, Bracarda S, Bukowski R, Catto J, Choueiri TK, Crabb S, Eisen T, El Demery M, Fitzpatrick J, Flamand V, Goebell PJ, Gravis G, Houede N, Jacqmin D, Kaplan R, Malavaud B, Massard C, Melichar B, Mourey L, Nathan P, Pasquier D, Porta C, Pouessel D, Quinn D, Ravaud A, Rolland F, Schmidinger M, Tombal B, Tosi D, Vauleon E, Volpe A, Wolter P, Escudier B, Filleron T; DATECAN Renal Cancer group. Guidelines for the definition of time-to-event end points in renal cell cancer clinical trials: results of the DATECAN projectdagger. Ann Oncol. 2015 Dec;26(12):2392-8. doi: 10.1093/annonc/mdv380. Epub 2015 Sep 14. PMID 26371288
- [Result] Cohen R, Vernerey D, Bellera C, Meurisse A, Henriques J, Paoletti X, Rousseau B, Alberts S, Aparicio T, Boukovinas I, Gill S, Goldberg RM, Grothey A, Hamaguchi T, Iveson T, Kerr R, Labianca R, Lonardi S, Meyerhardt J, Paul J, Punt CJA, Saltz L, Saunders MP, Schmoll HJ, Shah M, Sobrero A, Souglakos I, Taieb J, Takashima A, Wagner AD, Ychou M, Bonnetain F, Gourgou S, Yoshino T, Yothers G, de Gramont A, Shi Q, Andre T; ACCENT Group. Guidelines for time-to-event end-point definitions in adjuvant randomised trials for patients with localised colon cancer: Results of the DATECAN initiative. Eur J Cancer. 2020 May;130:63-71. doi: 10.1016/j.ejca.2020.02.009. Epub 2020 Mar 12. PMID 32172199

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sarcoma and GIST | Breast Cancer | Pancreatic Cancer | Renal Cell Carcinoma | Colon Cancer (Adjuvant Setting) | Solid Tumours Undergoing Image-guided Tumor Ablation | (Early) Non Small Cell Lung Cancer
Started | 32 | 35 | 33 | 36 | 24 | 36 | 69
Completed | 28 (Of the 32 experts who filled in the first questionnaire, 28 (87%) also participated in the second round of rating.) | 31 (Of the 35 experts who filled-in the first questionnaire, 31 (89%) also answered the second questionnaire.) | 30 (Of the 33 experts who filled-in the first questionnaire, 30 (91%) also answered the second questionnaire.) | 31 (Of the 36 experts who filled-in the first questionnaire, 31 (86%) also answered the second questionnaire.) | 24 (Of the 24 experts who completed the first questionnaire, 24 (100%) also answered the second round.) | 24 (Of the 36 experts who completed the first questionnaire, 24 (67%) also answered the second round.) | 54 (Of the 69 experts who filled in the first questionnaire, 54 (78%) also participated in the second round of rating.)
Not Completed | 4 | 4 | 3 | 5 | 0 | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sarcoma and GIST | Breast Cancer | Pancreatic Cancer | Renal Cell Carcinoma | Colon Cancer (Adjuvant Setting) | Solid Tumours Undergoing Image-guided Tumor Ablation | (Early) Non Small Cell Lung Cancer | Total
Number analyzed (Participants) | 28 | 31 | 30 | 31 | 24 | 24 | 54 | 222
Age, Customized [Count of Participants; unit: Participants] — Age of the medical experts who completed the survey questionnaire was not collected
  Participants
    18 years and older | 28 | 31 | 30 | 31 | 24 | 24 | 54 | 222
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 10 | 11 | 7 | 8 | 27 | 82
  Male | 20 | 20 | 20 | 20 | 17 | 16 | 27 | 140
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 6 | 15 | 17 | 11 | 3 | 1 | 8 | 61
  Italy | 4 | 1 | 2 | 3 | 3 | 1 | 8 | 22
  Denmark | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 4
  Belgium | 2 | 5 | 2 | 4 | 0 | 1 | 2 | 16
  United States | 6 | 0 | 0 | 3 | 6 | 5 | 9 | 29
  Netherlands | 3 | 2 | 1 | 2 | 1 | 5 | 7 | 21
  United Kingdom | 2 | 2 | 2 | 6 | 4 | 4 | 3 | 23
  Germany | 2 | 0 | 2 | 1 | 1 | 5 | 0 | 11
  Poland | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Portugal | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
  Slovenia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Greece | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3
  Spain | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Austria | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Canada | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Japan | 0 | 0 | 0 | 0 | 2 | 1 | 6 | 9
  Switzerland | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
  Australia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Argentina | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
  India | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Outcomes Defined Following the Consensus Process
Description: Number of time-to-event outcomes defined following the consensus process
Time Frame: 1 year after the consitution of the panel of experts
Population: For example: the 28 experts of the consensus panel involved in providing guidelines for time-to-event outcomes in Sarcoma and GIST trials provided recommandations for the definitions of 12 time to event outcomes to be used in randomized trials for sarcomas and GISTs. The precise definition of each outcome can be found in the publications.
Measure: Number; unit: Time to event outcomes
Arm/Group | Sarcoma and GIST | Breast Cancer | Pancreatic Cancer | Renal Cell Carcinoma | Colon Cancer (Adjuvant Setting) | Solid Tumours Undergoing Image-guided Tumor Ablation | (Early) Non Small Cell Lung Cancer
Number analyzed (Participants) | 28 | 31 | 33 | 36 | 24 | 36 | 54
Time to event outcomes | 12 | 11 | 14 | 7 | 5 | 4 | 19

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- (Early) Non Small Cell Lung Cancer: (early) Non Small Cell Lung Cancer : No intervention : Consensus of international experts to provide definition of survival endpoints to be used in randomized controlled trials to assess treatment efficacy.
Arm/Group | Sarcoma and GIST | Breast Cancer | Pancreatic Cancer | Renal Cell Carcinoma | Colon Cancer (Adjuvant Setting) | Solid Tumours Undergoing Image-guided Tumor Ablation | (Early) Non Small Cell Lung Cancer
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No